CLINICAL TRIAL: NCT05231330
Title: Clinical Evaluation of Silver Nanoparticles in Comparison to Silver Diamine Fluoride in Management of Deep Carious Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Kareem Hamdy Ahmed Aly, principal investigator, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR1
Record Dates: First submitted 2021-12-23; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- silver nanoparticles (Experimental)
  Interventions: Drug: silvernanoparticles
- silverdiamine fluoride (Active Comparator)
  Interventions: Drug: SDF
- no medicament (No Intervention)

INTERVENTIONS:
Drug: silvernanoparticles — silvernanoparticles in fluoride varnish
  Arms: silver nanoparticles
Drug: SDF — silver diamine fluoride
  Other Names: silver diamine fluoride
  Arms: silverdiamine fluoride

SUMMARY:
this clinical study will be carried out to evaluate the effect of fluoride varnish with silver nanoparticles in comparison to silver diamine fluoride in management of deep carious lesions.

ELIGIBILITY:
Inclusion Criteria:

* success will be evaluated by:

  1. Cold pulp testing: An ice-rod will be used for this test. Results should be positive or negative.
  2. Absence of spontaneous pain: Post-operative pain will be assessed using the visual Analogue Scale Score (VAS), which is a measurement method for subjective characteristics of pain. Respondents specify their level of agreement to a statement by indicating a position along a 10 cm line between two end-points, with the term "no sensitivity" at one end and "intolerable sensitivity" at the other end. A score from (0 to 10 is given).
  3. Sensitivity to percussion: (presence/ absence).
  4. Inspection for Sinus/fistula/swelling: using visual inspection (presence/ absence).
  5. Radiographic examination: Indicating presence of periapical radiolucencies, widening of lamina dura, internal and external root resorption (presence/ absence).

Exclusion Criteria:

* Patient-related criteria:

  * Medically compromised patients, who will not be able to attend multiple appointments or may require special management.
  * Pregnant women; as radiographs cannot be taken for them.
  * Allergy to any of the restorative materials, including anesthetics.
  * Uncooperative patients, will not abide by the instructions or attend the appointments.

Tooth related criteria:

* Retained deciduous teeth; as the study is targeting only permanent teeth.
* Teeth with previous restorations, which may add another variable to the study (type of old restorative material, extent of recurrent caries.
* Teeth with cervical caries; which can't be evaluated on periapical radiographs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Cold pulp testing | 6 months
  : An ice-rod will be used for this test. Results should be positive or negative.
Absence of spontaneous pain | 6 month
  Post-operative pain will be assessed using the visual Analogue Scale Score (VAS), which is a measurement method for subjective characteristics of pain. Respondents specify their level of agreement to a statement by indicating a position along a 10 cm line between two end-points, with the term "no sensitivity" at one end and "intolerable sensitivity" at the other end. A score from (0 to 10 is given).
Radiographic examination | 6 month
  Indicating presence of periapical radiolucencies, widening of lamina dura, internal and external root resorption (presence/ absence).
sensitivity to percussion | 6 month
  recorded as yes or no
visual inspection for sinus/ fistula swelling | 6 month
  recorded as yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Suez canal university, Suez, Egypt

IPD SHARING:
Plan to Share IPD: No